CLINICAL TRIAL: NCT05821647
Title: Effect of a Machine Learning-Derived Early Warning System for Hypotension vs Standard Care on Depth and Duration of Intra- and Postoperative Hypotension in Elective Cardiac Surgery
Brief Title: Hypotension Prediction 2 Study in Cardiac Surgery and Postoperative ICU Admission
Acronym: HYPE-2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Collaborators: Edwards Lifesciences (Industry)
Responsible Party: Principal Investigator, A.P.J. Vlaar, professor, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: NL76236.018.21; NL9449 (Registry Identifier: Netherlands Trial Registry)
Record Dates: First submitted 2023-02-28; First posted 2023-04-20 (Actual); Last update posted 2023-04-20 (Actual); Status verified 2023-04

CONDITIONS: Intraoperative Hypotension; Postoperative Hypotension; Hypotension
Keywords: Intensive Care Unit; Cardiac surgery; Coronary Artery Bypass Grafting
MeSH Terms: conditions — Hypotension

STUDY DESIGN:
Intervention Model Description: The study has two arms in which patients are allocated in a 1:1 randomization ratio.
Who Masked: Participant
Masking Description: The patient and the researcher performing the analysis are blinded. Because of the nature of the interventions, the investigators and treating anesthesiologist, anaesthesia nurse, intensivist and critical care nurse will not be masked to group allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): Objective to maintain a mean arterial blood pressure (MAP) above or equal to 65 mm Hg, as is standard care in out institution.
  This is done using standard hemodynamic monitoring, which in our center consists of continuous arterial blood pressure monitoring and the pulse pressure variation parameter. The clinician will administer either fluids, inotropes, vasopressors, or a combination, or apply positional changes to maintain the set MAP threshold.
- Additional HPI guided treatment (Experimental): Objective to maintain a mean arterial blood pressure (MAP) above or equal to 65 mm Hg, as is standard care in out institution.
  This is done using standard hemodynamic monitoring (as described for the control group) but is assisted by the Hypotension Prediction Index (HPI). This parameter is made available to the clinicians with the HemoSphere Advanced Monitoring Platform (HemoSphere) and is used to initiate treatment when the HPI values is ≥ 75.
  It also provides additional advanced hemodynamic variables (e.g. cardiac output, systemic vascular resistance). The treating clinicians are trained to use these variables and are provided with a diagnostic flowchart to determine the cause (preload, contractility and afterload) of the upcoming hypotensive (MAP < 65 mmHg) event. Timing of treatment and choice of treatment is then left to the discretion of the attending clinician.
  Interventions: Other: HPI guided treatment advice

INTERVENTIONS:
Other: HPI guided treatment advice — Administer hemodynamic altering intervention aimed at either a preload, contractility, or afterload problem to prevent impending hypotension. Treatment options include: administering either fluids, inotropes, vasopressors, positional changes, or a combination.
  Arms: Additional HPI guided treatment

SUMMARY:
This trial registration serves as an amendment incorporating the IPD Sharing Statement.

This study already has a trial registration (2021 April 30) in the Netherlands Trial Registry (Reference number NL9449, https://trialsearch.who.int/). However, the NTR register is subject to a merger with another Dutch register. This means that existing registrations are still visible, but can no longer be adjusted.

Study summary:

Hypotension in the operating room (OR) and during post-operative ICU admission is common in surgical patients and even more prevalent in cardiac surgery patients. It is associated with adverse outcomes and while these events are preventable, current management is predominantly reactive. Edwards Lifesciences (Irvine, CA) has developed the Hypotension Prediction Index (HPI), an early warning system that predicts an hypotensive event, defined as MAP below 65 mmHg, with high accuracy minutes before it occurs. At the time of writing the protocol this model has not been tested in a clinical trial in cardiac surgery patients or ICU admitted patients. The aim of the HYPE-2 trial is to assess whether the HPI-algorithm can reduce the time-weighted average (TWA) of intra- and postoperative hypotension in elective on-pump coronary artery bypass graft (CABG) surgery patients.

DETAILED DESCRIPTION:
Population studied:

All adult patients undergoing elective on-pump CABG surgery or CABG with additional single heart valve surgery (e.g. valve repair or replacement), requiring a radial arterial line and an intended target MAP of 65 mmHg or above during both surgery (excluding cardiopulmonary bypass pump time (CBP)) and during mechanically ventilated phase of duration of ICU admission.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older at inclusion
* Planned for elective on-pump CABG surgery or CABG with additional single heart valve surgery (e.g. valve repair or replacement)
* Planned to receive standard monitoring for cardiac surgery
* Target MAP of 65 mmHg or above during surgery
* Target MAP of 65 mmHg or above during the mechanically ventilated phase of ICU admission

Exclusion Criteria:

* Known cardiac shunts (significant)
* Severe cardiac arrhythmias (including but not limited to persistent atrial fibrillation prior to surgery)
* Expected to receive an hemodynamic assist device (e.g. intra-aortic balloon pump) during surgery
* Dialysis dependent kidney failure prior to surgery
* Planned to receive Perioperative Goal Directed Therapy (PGDT) other than standard intraoperative care
* Previous cardiac surgery in medical history

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2021-05-20 (Actual); Primary Completion 2023-02-16 (Actual); Study Completion 2023-03-16 (Actual)

PRIMARY OUTCOMES:
The overall time-weighted average (TWA) of hypotension (severity of hypotension) | During both the off-pump phases of on-pump CABG surgery and the mechanically ventilated phase of post-operative ICU admission (or 8 hours maximum)
  TWA is a calculation of the depth (in mmHg) of hypotension below the 'threshold' MAP of 65 mmHg x the time spent in hypotension in minutes, this resulting in an 'area'. To better compare this value between different patients the 'area' can be divided by the total duration of the measurement.

SECONDARY OUTCOMES:
Incidence of hypotension | Will be analyzed for the overall duration of both the off-pump phases of on-pump CABG surgery and the mechanically ventilated phase of post-operative ICU admission (or 8 hours maximum)
  number of hypotensive events during study phases
Time spent in hypotension | Will be analyzed for the overall duration of both the off-pump phases of on-pump CABG surgery and the mechanically ventilated phase of post-operative ICU admission (or 8 hours maximum)
  amount of time in minutes spent in hypotension during study phases
The percentage of time in hypotension | Will be analyzed for the overall duration of both the off-pump phases of on-pump CABG surgery and the mechanically ventilated phase of post-operative ICU admission (or 8 hours maximum)
  amount of time in hypotension expressed in percentage of the total study phases' duration
The AUT of a MAP < 65 mmHg | Will be analyzed for the overall duration of both the off-pump phases of on-pump CABG surgery and the mechanically ventilated phase of post-operative ICU admission (or 8 hours maximum)
  AUT is a calculation of the depth (in mmHg) of hypotension below the 'threshold' MAP of 65 mmHg x the time spent in hypotension in minutes, this resulting in an 'area'.
Incidence of hypertension | Will be analyzed for the overall duration of both the off-pump phases of on-pump CABG surgery and the mechanically ventilated phase of post-operative ICU admission (or 8 hours maximum)
  number of hypertensive events during study phases
Time spent in hypertension | Will be analyzed for the overall duration of both the off-pump phases of on-pump CABG surgery and the mechanically ventilated phase of post-operative ICU admission (or 8 hours maximum)
  amount of time in minutes spent in hypertension during study phases
The percentage of time in hypertension | Will be analyzed for the overall duration of both the off-pump phases of on-pump CABG surgery and the mechanically ventilated phase of post-operative ICU admission (or 8 hours maximum)
  amount of time in hypertension expressed in percentage of the total study phases' duration
The AAT of a MAP > 100 mmHg | Will be analyzed for the overall duration of both the off-pump phases of on-pump CABG surgery and the mechanically ventilated phase of post-operative ICU admission (or 8 hours maximum)
  AAT is a calculation of the depth (in mmHg) of hypertension above the 'threshold' MAP of 100 mmHg x the time spent in hypertension in minutes, this resulting in an 'area'.
TWA of hypertension | Will be analyzed for the overall duration of both the off-pump phases of on-pump CABG surgery and the mechanically ventilated phase of post-operative ICU admission (or 8 hours maximum)
  TWA is a calculation of the depth (in mmHg) of hypertension above the 'threshold' MAP of 100 mmHg x the time spent in hypertension in minutes, this resulting in an 'area'. This 'area' is divided by the total duration of the measurement.
Incidence of HPI alarm (HPI ≥ 75) | Will be analyzed for the overall duration of both the off-pump phases of on-pump CABG surgery and the mechanically ventilated phase of post-operative ICU admission (or 8 hours maximum)
  number of HPI alarms during study phases
Time spent in HPI alarm | Will be analyzed for the overall duration of both the off-pump phases of on-pump CABG surgery and the mechanically ventilated phase of post-operative ICU admission (or 8 hours maximum)
  amount of time in minutes spent in HPI alarms during study phases
The percentage of time in HPI alarm | Will be analyzed for the overall duration of both the off-pump phases of on-pump CABG surgery and the mechanically ventilated phase of post-operative ICU admission (or 8 hours maximum)
  amount of time in HPI alarms expressed in percentage of the total study phases' duration
The AAT of a HPI ≥ 75 | Will be analyzed for the overall duration of both the off-pump phases of on-pump CABG surgery and the mechanically ventilated phase of post-operative ICU admission (or 8 hours maximum)
  AAT is a calculation of the depth of HPI above or equal to the 'threshold' of 75 x the time spent in HPI alarm in minutes, this resulting in an 'area'.
TWA of HPI alarm | Will be analyzed for the overall duration of both the off-pump phases of on-pump CABG surgery and the mechanically ventilated phase of post-operative ICU admission (or 8 hours maximum)
  TWA is a calculation of the depth of HPI above or equal to the 'threshold' of 75 x the time spent in HPI alarm in minutes, this resulting in an 'area'. This 'area' is divided by the total duration of the measurement.
Treatment choice | Will be analyzed for the overall duration of both the off-pump phases of on-pump CABG surgery and the mechanically ventilated phase of post-operative ICU admission (or 8 hours maximum)
  vasopressors, blood transfusions, fluids, inotropes, position changes, decrease in anesthetics
Treatment dose | Will be analyzed for the overall duration of both the off-pump phases of on-pump CABG surgery and the mechanically ventilated phase of post-operative ICU admission (or 8 hours maximum)
  Dosage of medication or volume of fluids
Time to treatment | Will be analyzed for the overall duration of both the off-pump phases of on-pump CABG surgery and the mechanically ventilated phase of post-operative ICU admission (or 8 hours maximum)
  If an alarm or hypotensive event had more than 1 treatment, the time to first treatment will be used.
Number of treatments | Will be analyzed for the overall duration of both the off-pump phases of on-pump CABG surgery and the mechanically ventilated phase of post-operative ICU admission (or 8 hours maximum)
  amount of treatments (e.g., administered fluids, vasopressors, inotropes, anesthetics) given to alter the hemodynamics (increase of reduce the blood pressure)

OTHER OUTCOMES:
Incidence of hypertension (intraoperative) | During both the off-pump phases of on-pump CABG surgery (or 8 hours maximum)
  number of hypertensive events during the intraoperative study phases
Incidence of hypertension (postoperative in the ICU) | During the mechanically ventilated phase of post-operative ICU admission (or 8 hours maximum)
  number of hypertensive events during the ICU study phase
Time spent in hypertension (intraoperative) | During both the off-pump phases of on-pump CABG surgery (or 8 hours maximum)
  amount of time in minutes spent in hypertension during the intraoperative study phases
Time spent in hypertension (postoperative in the ICU) | During the mechanically ventilated phase of post-operative ICU admission (or 8 hours maximum)
  amount of time in minutes spent in hypertension during the ICU study phase
TWA of hypertension (intraoperative) | During both the off-pump phases of on-pump CABG surgery (or 8 hours maximum)
  TWA is a calculation of the depth (in mmHg) of hypertension above the 'threshold' MAP of 100 mmHg x the time spent in hypertension in minutes, this resulting in an 'area'. This 'area' is divided by the total duration of the measurement.
TWA of hypertension (postoperative in the ICU) | During the mechanically ventilated phase of post-operative ICU admission (or 8 hours maximum)
  TWA is a calculation of the depth (in mmHg) of hypertension above the 'threshold' MAP of 100 mmHg x the time spent in hypertension in minutes, this resulting in an 'area'. This 'area' is divided by the total duration of the measurement.
Incidence of HPI alarm (HPI ≥ 75) (intraoperative) | During both the off-pump phases of on-pump CABG surgery (or 8 hours maximum)
  number of HPI alarms during the intraoperative study phases
Incidence of HPI alarm (HPI ≥ 75) (postoperative in the ICU) | During the mechanically ventilated phase of post-operative ICU admission (or 8 hours maximum)
  number of HPI alarms during the ICU study phase
Time spent in HPI alarm (intraoperative) | During both the off-pump phases of on-pump CABG surgery (up to 8 hours)
  amount of time in minutes spent in HPI alarms during the intraoperative study phases
Time spent in HPI alarm (postoperative in the ICU) | During the mechanically ventilated phase of post-operative ICU admission (or 8 hours maximum)
  amount of time in minutes spent in HPI alarms during the ICU study phase
TWA of HPI alarm (intraoperative) | During both the off-pump phases of on-pump CABG surgery (or 8 hours maximum)
  TWA is a calculation of the depth of HPI above or equal to the 'threshold' of 75 x the time spent in HPI alarm in minutes, this resulting in an 'area'. This 'area' is divided by the total duration of the measurement.
TWA of HPI alarm (postoperative in the ICU) | During the mechanically ventilated phase of post-operative ICU admission (or 8 hours maximum)
  TWA is a calculation of the depth of HPI above or equal to the 'threshold' of 75 x the time spent in HPI alarm in minutes, this resulting in an 'area'. This 'area' is divided by the total duration of the measurement.
Compliance of clinicians to HPI treatment protocol + diagnostic guidance | Will be analyzed for all study phases of both the off-pump phases of on-pump CABG surgery and the mechanically ventilated phase of post-operative ICU admission (or 8 hours maximum)
  Assessed by the number of- and reason for protocol deviations: ignored treatment advices.
  The nurse driven hypotension treatment protocol only applies to the ICU nurses
Association between decrease in TWA of hypotension and a difference in creatinine (μmol/L) | Admission at ICU admission, and every morning of hospitalization after surgery (up to 28 days)
  Difference in laboratory value of creatinine between the control and HPI guided treatment group after the surgical procedure
Association between decrease in TWA of hypotension and a difference in lactate (mmol/L) | All lactate samples taken during the study phases and the samples taken every morning during ICU admission (up to 28 days)
  Difference in laboratory value of lactate between the control and HPI guided treatment group
Association between decrease in TWA of hypotension and a difference in creatinine kinase MB (μg/L) | During ICU admission (up to 28 days)
  Difference in laboratory value of creatinine kinase MB between the control and HPI guided treatment group
Association between decrease in TWA of hypotension and a difference in hematocrit (L/L) | During ICU admission (up to 28 days)
  Difference in laboratory value of hematocrit between the control and HPI guided treatment group
Association between decrease in TWA of hypotension and a difference in central venous oxygen saturation (%) | All samples taken during the study phases until the first sample after extubation at ICU (up to 28 days)
  Difference in laboratory value of central venous oxygen saturation between the control and HPI guided treatment group
Association between decrease in TWA of hypotension and a difference in brain natriuretic peptide (ng/L) | During ICU admission (up to 28 days)
  Difference in laboratory value of brain natriuretic peptide between the control and HPI guided treatment group
Sustained effect on TWA of hypotension | After HPI and diagnostic guidance is disconnected up to 8 hours after discontinuation.
  To study whether reducing the severity of hypotension with HPI and diagnostic guidance during both the surgery and the first hours of ICU admission results in a sustained effect after discontinuation of the HPI guided treatment.
Sustained effect on incidence of hypotension | After HPI and diagnostic guidance is disconnected up to 8 hours after discontinuation.
  To study whether reducing the severity of hypotension with HPI and diagnostic guidance during both the surgery and the first hours of ICU admission results in a sustained effect after discontinuation of the HPI guided treatment.
Sustained effect on time spent in hypotension | After HPI and diagnostic guidance is disconnected up to 8 hours after discontinuation.
  To study whether reducing the severity of hypotension with HPI and diagnostic guidance during both the surgery and the first hours of ICU admission results in a sustained effect after discontinuation of the HPI guided treatment.
Difference in treatment behaviour between groups expressed as total number of alarms (n) | Will be analyzed for all study phases of both the off-pump phases of on-pump CABG surgery and the mechanically ventilated phase of post-operative ICU admission (or 8 hours maximum)
  To study control group's treatment behaviour after silent alarms to which they were blinded and compare this with treatment behaviour after alarms in the HPI guided treatment group. This analysis focusses on the number of treatments after an early warning system alarm (referred to as 'alarm') but before hypotension occurred. In the HPI guided treatment group the alarms were visible to the treating anesthesiologists. In the control group the alarms were not visible to the treating anesthesiologists. The researchers will compare the total number of alarms (n) between both groups.
Difference in treatment behaviour between groups expressed as number of alarms per patients (n) | Will be analyzed for all study phases of both the off-pump phases of on-pump CABG surgery and the mechanically ventilated phase of post-operative ICU admission (or 8 hours maximum)
  To study control group's treatment behaviour after silent alarms to which they were blinded and compare this with treatment behaviour after alarms in the HPI guided treatment group. This analysis focusses on the number of treatments after an early warning system alarm (referred to as 'alarm') but before hypotension occurred. In the HPI guided treatment group the alarms were visible to the treating anesthesiologists. In the control group the alarms were not visible to the treating anesthesiologists. The researchers will compare the number of alarms per patients (n) between both groups.
Difference in treatment behaviour between groups expressed as total percentage of alarms treated (%) | Will be analyzed for all study phases of both the off-pump phases of on-pump CABG surgery and the mechanically ventilated phase of post-operative ICU admission (or 8 hours maximum)
  To study control group's treatment behaviour after silent alarms to which they were blinded and compare this with treatment behaviour after alarms in the HPI guided treatment group. This analysis focusses on the number of treatments after an early warning system alarm (referred to as 'alarm') but before hypotension occurred. In the HPI guided treatment group the alarms were visible to the treating anesthesiologists. In the control group the alarms were not visible to the treating anesthesiologists. The researchers will compare the total percentage of alarms treated (%) for each group.
Difference in treatment behaviour between groups expressed as time from alarm to first treatment action (seconds). | Will be analyzed for all study phases of both the off-pump phases of on-pump CABG surgery and the mechanically ventilated phase of post-operative ICU admission (or 8 hours maximum)
  To study control group's treatment behaviour after silent alarms to which they were blinded and compare this with treatment behaviour after alarms in the HPI guided treatment group. This analysis focusses on the number of treatments after an early warning system alarm (referred to as 'alarm') but before hypotension occurred. In the HPI guided treatment group the alarms were visible to the treating anesthesiologists. In the control group the alarms were not visible to the treating anesthesiologists. The researchers will compare the time from alarm occurrences to first treatment action (seconds).
Difference in treatment behaviour between groups expressed as time from first alarm to first treatment action (seconds). | Will be analyzed for all study phases of both the off-pump phases of on-pump CABG surgery and the mechanically ventilated phase of post-operative ICU admission (or 8 hours maximum)
  To study control group's treatment behaviour after silent alarms to which they were blinded and compare this with treatment behaviour after alarms in the HPI guided treatment group. This analysis focusses on the number of treatments after an early warning system alarm (referred to as 'alarm') but before hypotension occurred. In the HPI guided treatment group the alarms were visible to the treating anesthesiologists. In the control group the alarms were not visible to the treating anesthesiologists. The researchers will compare the time from first alarm to first treatment action (seconds).
Assess required treatment during hypotension (MAP < 65 mmHg) within both off-pump phases of on-pump CABG surgery as the determined by the anesthesiologist based on transesophageal echocardiogram (TEE) observations. | During hemodynamic instability (hypotension) within both the off-pump phases of on-pump CABG surgery (or 8 hours maximum)
  Anesthesiologists have the expertise to use TEE observations during hypotensive events to obtain insight in the most likely cause of hypotension: hypovolemia, vasoplegia or reduced ventricular contractility. Each time these observations are obtained the researchers will annotate the determined required treatment.
Assess required treatment during hypotension (MAP < 65 mmHg) within both off-pump phases of on-pump CABG surgery as the determined by the diagnostic guidance protocol. | During hemodynamic instability (hypotension) within both the off-pump phases of on-pump CABG surgery (or 8 hours maximum)
  Prior to the start of the study the researchers designed a diagnostic guidance protocol that integrates parameters obtained from the HemoSphere monitor (i.e., stroke volume, stroke volume variation, systemic vascular resistance, and Dynamic arterial elastance). These parameters provide insight in the most likely cause of forthcoming hypotension: hypovolemia, vasoplegia or reduced ventricular contractility. During hemodynamic instability and hypotension the diagnostic guidance protocl is used to determine the required treatment and will be annotated.
Relation between required treatment as determined by the anesthesiologist's expertise using TEE observations versus the required treatment as determined using the diagnostic guidance protocol. | During hemodynamic instability within both the off-pump phases of on-pump CABG surgery (up to 8 hours)
  As described in the outcome measures 46 and 47, the researchers will assess the required treatments during hemodynamic instability and hypotension. These treatments are determined by the anesthesiologists using TEE observations and simultaneously also by the researchers using the study's diagnostic guidance protocol. Both diagnostic strategies will determine the same treatment options, namely: hypovolemia, vasoplegia or reduced ventricular contractility. The researchers will assess the number of devations in determined treatment.

CONTACTS AND LOCATIONS:
Overall Officials: A.P.J. Vlaar, Principal Investigator — Department of Intensive Care, Amsterdam UMC, location AMC, Amsterdam, the Netherlands
Locations (1):
- Amsterdam University Medical Centers, Amsterdam-Zuidoost, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in the final article including results in the text, tables, figures, and appendices, will be made available after deidentification.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: After 3 months and ending 36 months following article publication
Access Criteria: Researchers who provide a methodologically sound proposal to achieve results in line with the proposed outcomes will be able to obtain IPD.

REFERENCES:
- [Background] Wijnberge M, Geerts BF, Hol L, Lemmers N, Mulder MP, Berge P, Schenk J, Terwindt LE, Hollmann MW, Vlaar AP, Veelo DP. Effect of a Machine Learning-Derived Early Warning System for Intraoperative Hypotension vs Standard Care on Depth and Duration of Intraoperative Hypotension During Elective Noncardiac Surgery: The HYPE Randomized Clinical Trial. JAMA. 2020 Mar 17;323(11):1052-1060. doi: 10.1001/jama.2020.0592. PMID 32065827
- [Background] Hatib F, Jian Z, Buddi S, Lee C, Settels J, Sibert K, Rinehart J, Cannesson M. Machine-learning Algorithm to Predict Hypotension Based on High-fidelity Arterial Pressure Waveform Analysis. Anesthesiology. 2018 Oct;129(4):663-674. doi: 10.1097/ALN.0000000000002300. PMID 29894315
- [Derived] Schuurmans J, Rellum SR, Schenk J, van der Ster BJP, van der Ven WH, Geerts BF, Hollmann MW, Cherpanath TGV, Lagrand WK, Wynandts PR, Paulus F, Driessen AHG, Terwindt LE, Eberl S, Hermanns H, Veelo DP, Vlaar APJ. Effect of a Machine Learning-Derived Early Warning Tool With Treatment Protocol on Hypotension During Cardiac Surgery and ICU Stay: The Hypotension Prediction 2 (HYPE-2) Randomized Clinical Trial. Crit Care Med. 2025 Feb 1;53(2):e328-e340. doi: 10.1097/CCM.0000000000006518. Epub 2024 Nov 22. PMID 39576150
- [Derived] Rellum SR, Schuurmans J, Schenk J, van der Ster BJP, van der Ven WH, Geerts BF, Hollmann MW, Cherpanath TGV, Lagrand WK, Wynandts P, Paulus F, Driessen AHG, Terwindt LE, Eberl S, Hermanns H, Veelo DP, Vlaar APJ. Effect of the machine learning-derived Hypotension Prediction Index (HPI) combined with diagnostic guidance versus standard care on depth and duration of intraoperative and postoperative hypotension in elective cardiac surgery patients: HYPE-2 - study protocol of a randomised clinical trial. BMJ Open. 2023 May 2;13(5):e061832. doi: 10.1136/bmjopen-2022-061832. PMID 37130670